CLINICAL TRIAL: NCT02119455
Title: Biomarkers of Orthodontic Tooth Movement With Fixed Appliances and Vibration Appliance Therapy: A Randomized Clinical Trial
Brief Title: Biomarkers of Orthodontic Tooth Movement With Fixed Appliances and Vibration Appliance Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: OrthoAccel Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Taranpreet Chandhoke, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OATI-20130635
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Tooth Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vibration Device+Fixed Appliance Tx (Experimental): Male and female subjects will randomly assigned to this group to receive fixed appliance orthodontic treatment in conjunction with vibration therapy (daily use of OrthoAccel Aura device for 20 minutes/day) during the study period.
  Interventions: Device: Vibration Device
- No Vibration Device+Fixed Appliance Tx (No Intervention): Male and female subjects will randomly assigned to this group to receive fixed appliance orthodontic treatment only and no vibration treatment.

INTERVENTIONS:
Device: Vibration Device — Subjects receiving the OrthoAccel Aura device will be instructed to use the device for 20 minutes/day per the manufacturer's instructions during the study period.
  Arms: Vibration Device+Fixed Appliance Tx

SUMMARY:
Currently, orthodontic treatment typically lasts approximately 2 years. There are a number of advantages for reducing the duration of treatment, including reducing the potential risk of caries, root resorption and for minimizing patient "burn out" from prolonged treatment.

While some evidence does exist that vibration may accelerate the speed of tooth movement, the biological mechanism is still unknown. Identification of specific factors involved in tooth movement that are further stimulated by vibration would help to understand the mechanisms involved as well as discover possible biologic targets which could be utilized or modified to maximize the benefits of vibration treatment.

The purpose of this study is to identify novel biological factors that are expressed in patients undergoing orthodontic tooth movement in conjunction with vibration appliance therapy.

DETAILED DESCRIPTION:
Specific Aims

1. To determine if combined vibration-fixed appliance treatment alters the expression of specific bone remodeling factors in saliva compared to fixed orthodontic treatment alone.
2. To further elucidate the role of vibration treatment on the degree of tooth mobility during fixed appliance treatment compared to control.
3. To determine if combined vibration-fixed appliance treatment increases the speed of orthodontic tooth movement during the alignment phase of treatment.
4. To evaluate the role of vibration treatment in the control of pain in patients undergoing orthodontic treatment.

Screening & Recruitment Procedures Approximately 600 patients begin treatment every year in the University of Connecticut Orthodontic Clinic. The pilot project aim is to recruit a total of 40 patients, with 20 male and 20 female subjects, equally divided between control and vibration groups. Based on the projected starts, we anticipate meeting the recruitment goals during the first 12 months of the study.

Prospective subjects will be screened for this study after completing all the usual initial screening procedures for patients in the University of Connecticut Orthodontic Clinic with their appointed primary orthodontic provider. The primary orthodontic provider will determine if the patient is likely to qualify (pre-screen) for the study based on the inclusion/exclusion criteria. The initial clinical indicators of eligibility evaluated during the pre-screen are a healthy patient undergoing non-extraction treatment with good oral hygiene. Male and female subjects of all ethnicities will be included if between the ages of 15-35 years of age.

If the prospective patient meets the initial criteria, the orthodontic provider will notify the study coordinator and PI to screen the patient's existing dental records, including screening forms, models and/or radiographs for confirmation of likely eligibility for participation in the study.

Study Procedures I. Standardized Orthodontic Treatment Protocol The orthodontic clinic treatment protocol will be standardized to minimize variability in the sequence of treatment. All subjects will be bonded with 0.022"X0.028" brackets passive self-ligating brackets with maximal band tension (MBT) prescription from 2nd premolar to 2nd premolar in both arches and bonded tubes on the 1st molars at the baseline (T0) visit. Each subject will have a 0.014" copper nickel titanium (NiTi) archwire placed at the initial visit. At T2, the next archwire in the sequence (0.014"X0.025" copper NiTi) will be placed.

Subjects will be seen at normally appointed visits every 4-6 weeks. The primary orthodontic provider will direct the alignment and leveling phase of treatment and proceed through the wire sequence as indicated. No specific procedure/timeframe will be assigned to placement of each archwire. Providers are expected to proceed to the next archwire when it can be placed comfortably based on the degree of alignment achieved.

In the event of bracket breakages, the subject is to be seen within 7 days to have the bracket rebonded, in standard care as well as the study. The primary orthodontic provider will reposition the bracket in the ideal position and continue with alignment using the study archwires. If the subject does not present with 7 days of the breakage, he/she will be disqualified from the study.

II. Randomization Procedures Once recruited to the study and after baseline measures are taken at T0 by the study coordinator, the randomization will be performed. Since study groups will be subdivided by gender, separate randomization will be performed for males and females. Block randomization will be used. Based on gender, 20 opaque envelopes will be generated containing the group allocation (10 for the vibration study group, 10 for the non-vibration control group). At the time of randomization, the subject will choose an envelope and disclose the group assignment. For subjects allocated to the vibration group, the study coordinator will provide detailed instructions as to how to operate the appliance and will instruct those subjects to use it for 20 minutes per day.

III. Data Collection Procedures On the day of bonding (T0), prior to the placement of any appliances, baseline unstimulated whole saliva will be collected and Periotest will performed on selected teeth in the mandibular arch. In addition, alginate model impressions will be taken. These procedures will be described in more detail in the next sections. Once baseline measures have been taken, the PI will perform the randomization and notify the study coordinator as to which group the subject is assigned to ("vibration treatment" or "no vibration"). The patients allocated to the vibration treatment group will be provided with the vibration appliance (Acceledent) appliance and instructed to use the 20 minutes per day according to the manufacturer's instructions.

After fixed appliances are placed and tooth movement begins, subjects will proceed with standard orthodontic treatment with or without vibration treatment based on allocation. Collection of saliva samples, Periotest and alginate impressions will be taken at T1 (5-6 weeks post-T0), T2 (10-12 weeks post-T0) and T3 (15-17 weeks post-T0). Subjects will be seen between noon and 5pm to help minimize possible confounding of salivary markers by circadian rhythms.

Salivary Biomarkers Collection of unstimulated whole saliva will be performed using the same methods described by Navazesh and Kumar. Unstimulated whole saliva will be collected by passive drooling into sterile centrifuge tubes on ice for 15 minutes or once 2-10 milliliters (mL) of saliva is collected at baseline and each visit, whichever occurs first. Once saliva is collected, samples will be kept on ice and supplemented with proteinase inhibitor. Samples will then be centrifuged for 10 minutes at 3000 rpm to remove cellular debris and supernatants will be collected and stored at -80°C until they are ready to be analyzed for biomarkers.

Biomarkers will be evaluated by ELISA assay by a direct sandwich method using a standard protocol.

Periotest Measurement Procedures This measurement is obtained at baseline and each visit. The degree of tooth mobility will be used using a Periotest device (Siemens, Bensheim, Germany) on the central incisors, canines and 2nd premolars in both mandibular quadrants as previously described by Liou et al. The archwire will be removed and the Periotest measurements will be taken in triplicate, with means recorded.

Dental Model Analysis

Two blinded clinical evaluators will assess the rate of alignment of the lower incisors for both groups. Analyses of dental casts will be done on the mandibular cast using a method based on Little's irregularity index. Little's irregularity index was developed to assess amount of anterior tooth displacement from canine to canine. Contact displacement will be measured in millimeters around the arch from canine to canine. Irregularity will be measured on models from each of the four time points and be evaluated based on percentage change over the 6-month evaluation period.

Orthodontic Pain Assessment

Subjects will be given a pain diary on the baseline (T0), visits T1 & T2 to record the level of orthodontic pain each evening for the first 7 days after each study visit. The degree of pain will be assessed using a Visual Analog Scale (VAS) ranging from 1 (least pain) to 10 (highest pain). In addition, patients will report if the pain is constant or only present on biting/chewing. The subjects will return the completed diary to the next visit to be collected by the study coordinator and kept in the study record.

Oral Health Quality of Life (OHQoL)

To assess the impact of the vibration appliance on the overall oral health quality of life of the subject, subjects will be given an Oral Health Impact Profile (OHIP-14) questionnaire. The OHIP-14 consists of 14 questions divided into specific dimensions including functional limitation, physical pain, psychological discomfort, physical disability, psychological and social disability and overall life handicap from orthodontic treatment with or without the vibration appliance. The OHIP-14 will be administered at each study visit and the profile changes will be compared across time points in data analyses.

Individual scores are multiplied by the weights to give a subscale score for each category.

IV. Sample size and justification Few studies exist evaluating salivary biomarkers during orthodontic tooth movement. Our primary outcome is changes in the expression of specific biomarkers of cellular activation and bone remodeling. No randomized clinical trials (RCTs) are currently available to predict treatment effects on biomarker expression. This study will serve as a pilot project with 40 patients total in 4 groups divided by gender and vibration/no-vibration treatment arms.

We estimate 600 patients in the target age range beginning orthodontic treatment at the University of Connecticut Orthodontic Clinic each year. We anticipate meeting our recruitment goal for this study.

V. Subject Participation The timing of visit activity is planned to coincide with normally scheduled clinic provider/patient visits. Typically, treatment for non-extraction cases last from 12-30 months in the Orthodontic clinic using fixed appliances. However, the subjects will only be evaluated during the first 6 months of their clinical appliance treatment for the study purpose and data. Providers will follow patients every 5-6 weeks and the study coordinator will ensure/confirm the patients for study appointments. After completion of the observation and data collection phase ( up to 17 weeks), the patients will continue to proceed with treatment as directed by the their primary orthodontic provider. Data collection will occur at normally scheduled visits with no additional appointments specific to the study.

In the event that the PI determines that a subject is not suited to continue in the study (eg. the subject shows consistent failure to keep appointed visits, consistent breakage of appliances, patient safety considerations, etc.) he/she will be withdrawn by the PI from the study and no further data will be collected. Specifically, poor compliance with attending appointments during the allotted time frame for each study visit will result in subjects being disqualified from the study. For example, the follow-up time frame for T1 is 5-6 weeks after T0 (baseline). Therefore if the patient misses an appointment and cannot or does not reschedule to attend his/her appoint during the allotted time from (by 6 weeks after T0), then he/she will be disqualified from the study. Also, in the event of bracket breakages (as stated earlier), the subject is to be seen within 7 days to have the bracket rebounded. The primary orthodontic provider will reposition the bracket in the ideal position and continue with alignment using the study archwires. If the subject does not present with 7 days of the breakage, he/she will be disqualified from the study.

The data collected to that point will be utilized in analyses. The patient's treatment will continue with the primary orthodontic provider consistent with the standard of care.

VI. Statistical/Data Analysis Intra and inter-rater reliability of the irregularity measurements will be assessed using the T0 and T3 models evaluated by the two blinded evaluators one week apart for all patients. A Cronbach alpha analysis will be used to assess reliability of the measurements. A single calibrated evaluator (the study coordinator) will collect all tooth mobility measurements with the Periotest and means will be evaluated using non-parametric statistical analyses.

A Wilcoxon Rank Sum test for independent samples will be used to assess differences between groups for all the continuous variables with an α=0.05 for irregularity index changes-Periotest measurements, VAS &OHIP-14 measures.

Salivary biomarker expression will be analyzed by ANOVA to assess differences between the four study groups at each time point. The study coordinator and principal investigator will perform statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoker with no systemic medical conditions and no routine medications
* 15 to 35 years of age at the time of bonding
* Non-extraction treatment plan or no extractions required in the first 6 months of treatment
* At least 5mm of crowding in the mandibular arch
* Full-complement dentition 1st molar to 1st molar
* Good oral hygiene

Exclusion Criteria:

* Patients that require extractions as part of the orthodontic plan
* Smoking or excessive alcohol consumption
* Patients with edentulous areas
* Evidence of periodontal disease (any pocket depths more than 4mm)
* Use of anti-inflammatory drugs within 2 days of bonding
* Active oral lesions (ulcerations, sores, mucositis, etc.)
* Uncontrolled diabetes
* Dentofacial deformities (cleft palate, hemifacial microsomia, etc.)
* Subjects routinely taking any of the following medications:
* Corticosteroids (including for asthma)
* Bisphosphonates
* Anti-inflammatories
* Nicotine Patch
* Estrogen
* Opioids
* Growth Hormone
* Relaxin
* Anti-coagulants
* Disease that could affect bone metabolism:
* Parathyroid or thyroid dysfunction
* Osteoporosis, osteomalacia
* Vitamin D deficiency
* Fibrous dysplasia
* Paget's Disease
* Multiple Myeloma
* Osteogenesis Imperfecta
* History of Bone Metastasis
* Patients taking medications such as bisphosphonates, corticosteroids or any anti-inflammatory drug

Ages: 15 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taranpreet K Chandhoke, DMD, PhD, Principal Investigator — UCHC Department of Craniofacial Sciences; Flavio A Uribe, DDS, MDentSc, Principal Investigator — UCHC Department of Craniofacial Sciences
Locations (1):
- University of Connecticut Division of Orthodontics, Farmington, Connecticut, United States

REFERENCES:
- [Background] Miricescu D, Totan A, Calenic B, Mocanu B, Didilescu A, Mohora M, Spinu T, Greabu M. Salivary biomarkers: relationship between oxidative stress and alveolar bone loss in chronic periodontitis. Acta Odontol Scand. 2014 Jan;72(1):42-7. doi: 10.3109/00016357.2013.795659. Epub 2013 Jul 22. PMID 23869629
- [Background] Zhang F, Wang CL, Koyama Y, Mitsui N, Shionome C, Sanuki R, Suzuki N, Mayahara K, Shimizu N, Maeno M. Compressive force stimulates the gene expression of IL-17s and their receptors in MC3T3-E1 cells. Connect Tissue Res. 2010 Oct;51(5):359-69. doi: 10.3109/03008200903456942. PMID 20497006
- [Background] Andrade I Jr, Silva TA, Silva GA, Teixeira AL, Teixeira MM. The role of tumor necrosis factor receptor type 1 in orthodontic tooth movement. J Dent Res. 2007 Nov;86(11):1089-94. doi: 10.1177/154405910708601113. PMID 17959902
- [Background] Asano M, Yamaguchi M, Nakajima R, Fujita S, Utsunomiya T, Yamamoto H, Kasai K. IL-8 and MCP-1 induced by excessive orthodontic force mediates odontoclastogenesis in periodontal tissues. Oral Dis. 2011 Jul;17(5):489-98. doi: 10.1111/j.1601-0825.2010.01780.x. Epub 2010 Dec 23. PMID 21496183
- [Background] Basaran G, Ozer T, Kaya FA, Kaplan A, Hamamci O. Interleukine-1beta and tumor necrosis factor-alpha levels in the human gingival sulcus during orthodontic treatment. Angle Orthod. 2006 Sep;76(5):830-6. doi: 10.1043/0003-3219(2006)076[0830:IATNFL]2.0.CO;2. PMID 17029518
- [Background] Bildt MM, Bloemen M, Kuijpers-Jagtman AM, Von den Hoff JW. Matrix metalloproteinases and tissue inhibitors of metalloproteinases in gingival crevicular fluid during orthodontic tooth movement. Eur J Orthod. 2009 Oct;31(5):529-35. doi: 10.1093/ejo/cjn127. Epub 2009 Mar 18. PMID 19299245
- [Background] Brosens V, Ghijselings I, Lemiere J, Fieuws S, Clijmans M, Willems G. Changes in oral health-related quality of life reports in children during orthodontic treatment and the possible role of self-esteem: a follow-up study. Eur J Orthod. 2014 Apr;36(2):186-91. doi: 10.1093/ejo/cjt035. Epub 2013 Jun 6. PMID 23744704
- [Background] Brudvik P, Rygh P. Root resorption after local injection of prostaglandin E2 during experimental tooth movement. Eur J Orthod. 1991 Aug;13(4):255-63. doi: 10.1093/ejo/13.4.255. PMID 1717297
- [Background] Canavarro C, Teles RP, Capelli Junior J. Matrix metalloproteinases -1, -2, -3, -7, -8, -12, and -13 in gingival crevicular fluid during orthodontic tooth movement: a longitudinal randomized split-mouth study. Eur J Orthod. 2013 Oct;35(5):652-8. doi: 10.1093/ejo/cjs053. Epub 2012 Sep 17. PMID 22989715
- [Background] Capelli J Jr, Kantarci A, Haffajee A, Teles RP, Fidel R Jr, Figueredo CM. Matrix metalloproteinases and chemokines in the gingival crevicular fluid during orthodontic tooth movement. Eur J Orthod. 2011 Dec;33(6):705-11. doi: 10.1093/ejo/cjq148. Epub 2011 Mar 9. PMID 21389074
- [Background] Darendeliler MA, Zea A, Shen G, Zoellner H. Effects of pulsed electromagnetic field vibration on tooth movement induced by magnetic and mechanical forces: a preliminary study. Aust Dent J. 2007 Dec;52(4):282-7. doi: 10.1111/j.1834-7819.2007.tb00503.x. PMID 18265683
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Feu D, Miguel JA, Celeste RK, Oliveira BH. Effect of orthodontic treatment on oral health-related quality of life. Angle Orthod. 2013 Sep;83(5):892-8. doi: 10.2319/100412-781.1. Epub 2013 Apr 17. PMID 23593976
- [Background] Grant M, Wilson J, Rock P, Chapple I. Induction of cytokines, MMP9, TIMPs, RANKL and OPG during orthodontic tooth movement. Eur J Orthod. 2013 Oct;35(5):644-51. doi: 10.1093/ejo/cjs057. Epub 2012 Sep 17. PMID 22987319
- [Background] Greabu M, Didilescu A, Puiu L, Miricescu D, Totan A. Salivary antioxidant biomarkers in non-ferrous metals mine workers--a pilot study. J Oral Pathol Med. 2012 Jul;41(6):490-3. doi: 10.1111/j.1600-0714.2012.01131.x. Epub 2012 Mar 7. PMID 22394326
- [Background] Henriksen K, Andersen JR, Riis BJ, Mehta N, Tavakkol R, Alexandersen P, Byrjalsen I, Valter I, Nedergaard BS, Teglbjaerg CS, Stern W, Sturmer A, Mitta S, Nino AJ, Fitzpatrick LA, Christiansen C, Karsdal MA. Evaluation of the efficacy, safety and pharmacokinetic profile of oral recombinant human parathyroid hormone [rhPTH(1-31)NH(2)] in postmenopausal women with osteoporosis. Bone. 2013 Mar;53(1):160-6. doi: 10.1016/j.bone.2012.11.045. Epub 2012 Dec 9. PMID 23234813
- [Background] Jacobs C, Walter C, Ziebart T, Grimm S, Meila D, Krieger E, Wehrbein H. Induction of IL-6 and MMP-8 in human periodontal fibroblasts by static tensile strain. Clin Oral Investig. 2014 Apr;18(3):901-8. doi: 10.1007/s00784-013-1032-1. Epub 2013 Jul 14. PMID 23851938
- [Background] John MT, Patrick DL, Slade GD. The German version of the Oral Health Impact Profile--translation and psychometric properties. Eur J Oral Sci. 2002 Dec;110(6):425-33. doi: 10.1034/j.1600-0722.2002.21363.x. PMID 12507215
- [Background] Jonsson A, Malmgren O, Levander E. Long-term follow-up of tooth mobility in maxillary incisors with orthodontically induced apical root resorption. Eur J Orthod. 2007 Oct;29(5):482-7. doi: 10.1093/ejo/cjm047. PMID 17974537
- [Background] Krishnan V, Davidovitch Z. The effect of drugs on orthodontic tooth movement. Orthod Craniofac Res. 2006 Nov;9(4):163-71. doi: 10.1111/j.1601-6343.2006.00372.x. PMID 17101023
- [Background] Krishnan V, Davidovitch Z. On a path to unfolding the biological mechanisms of orthodontic tooth movement. J Dent Res. 2009 Jul;88(7):597-608. doi: 10.1177/0022034509338914. PMID 19641146
- [Background] Kumar S, Ram S, Navazesh M. Salivary gland and associated complications in head and neck cancer therapy. J Calif Dent Assoc. 2011 Sep;39(9):639-47. PMID 22034798
- [Background] Lee TY, Lee KJ, Baik HS. Expression of IL-1beta, MMP-9 and TIMP-1 on the pressure side of gingiva under orthodontic loading. Angle Orthod. 2009 Jul;79(4):733-9. doi: 10.2319/031308-145.1. PMID 19537852
- [Background] Leonardi R, Talic NF, Loreto C. MMP-13 (collagenase 3) immunolocalisation during initial orthodontic tooth movement in rats. Acta Histochem. 2007;109(3):215-20. doi: 10.1016/j.acthis.2007.01.002. Epub 2007 Mar 9. PMID 17350083
- [Background] Liou EJ, Chen PH, Wang YC, Yu CC, Huang CS, Chen YR. Surgery-first accelerated orthognathic surgery: postoperative rapid orthodontic tooth movement. J Oral Maxillofac Surg. 2011 Mar;69(3):781-5. doi: 10.1016/j.joms.2010.10.035. PMID 21353934
- [Background] Liou EJ, Chen PH, Wang YC, Yu CC, Huang CS, Chen YR. Surgery-first accelerated orthognathic surgery: orthodontic guidelines and setup for model surgery. J Oral Maxillofac Surg. 2011 Mar;69(3):771-80. doi: 10.1016/j.joms.2010.11.011. Epub 2011 Jan 22. PMID 21257249
- [Background] Lisboa RA, Andrade MV, Cunha-Melo JR. Toll-like receptor activation and mechanical force stimulation promote the secretion of matrix metalloproteinases 1, 3 and 10 of human periodontal fibroblasts via p38, JNK and NF-kB. Arch Oral Biol. 2013 Jun;58(6):731-9. doi: 10.1016/j.archoralbio.2012.12.009. Epub 2013 Jan 14. PMID 23332208
- [Background] Locker D, Slade G. Oral health and the quality of life among older adults: the oral health impact profile. J Can Dent Assoc. 1993 Oct;59(10):830-3, 837-8, 844. PMID 8221283
- [Background] Lukas D, Schulte W, Konig M, Reim M. High-speed filming of the Periotest measurement. J Clin Periodontol. 1992 Jul;19(6):388-91. doi: 10.1111/j.1600-051x.1992.tb00667.x. PMID 1634628
- [Background] Madureira DF, Taddei Sde A, Abreu MH, Pretti H, Lages EM, da Silva TA. Kinetics of interleukin-6 and chemokine ligands 2 and 3 expression of periodontal tissues during orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2012 Oct;142(4):494-500. doi: 10.1016/j.ajodo.2012.05.012. PMID 22999673
- [Background] Miles P, Smith H, Weyant R, Rinchuse DJ. The effects of a vibrational appliance on tooth movement and patient discomfort: a prospective randomised clinical trial. Aust Orthod J. 2012 Nov;28(2):213-8. PMID 23304970
- [Background] Masini V. [Sexual activity after myocardial infarct]. G Ital Cardiol. 1980;10(3):241-5. No abstract available. Italian. PMID 7372039
- [Background] Mummolo S, Marchetti E, Giuca MR, Gallusi G, Tecco S, Gatto R, Marzo G. In-office bacteria test for a microbial monitoring during the conventional and self-ligating orthodontic treatment. Head Face Med. 2013 Feb 1;9:7. doi: 10.1186/1746-160X-9-7. PMID 23375053
- [Background] Nagase S, Hashimoto Y, Small M, Ohyama M, Kuwayama T, Deacon S. Serum and urine bone resorption markers and pharmacokinetics of the cathepsin K inhibitor ONO-5334 after ascending single doses in post menopausal women. Br J Clin Pharmacol. 2012 Dec;74(6):959-70. doi: 10.1111/j.1365-2125.2012.04307.x. PMID 22533981
- [Background] Nammontri O, Robinson PG, Baker SR. Enhancing oral health via sense of coherence: a cluster-randomized trial. J Dent Res. 2013 Jan;92(1):26-31. doi: 10.1177/0022034512459757. Epub 2012 Sep 27. PMID 23018820
- [Background] Nanitsos E, Vartuli R, Forte A, Dennison PJ, Peck CC. The effect of vibration on pain during local anaesthesia injections. Aust Dent J. 2009 Jun;54(2):94-100. doi: 10.1111/j.1834-7819.2009.01100.x. PMID 19473149
- [Background] Navazesh M, Kumar SK. Xerostomia: prevalence, diagnosis, and management. Compend Contin Educ Dent. 2009 Jul-Aug;30(6):326-8, 331-2; quiz 333-4. PMID 19715009
- [Background] Navazesh M, Kumar SK; University of Southern California School of Dentistry. Measuring salivary flow: challenges and opportunities. J Am Dent Assoc. 2008 May;139 Suppl:35S-40S. doi: 10.14219/jada.archive.2008.0353. PMID 18460678
- [Background] Nishimura M, Chiba M, Ohashi T, Sato M, Shimizu Y, Igarashi K, Mitani H. Periodontal tissue activation by vibration: intermittent stimulation by resonance vibration accelerates experimental tooth movement in rats. Am J Orthod Dentofacial Orthop. 2008 Apr;133(4):572-83. doi: 10.1016/j.ajodo.2006.01.046. PMID 18405822
- [Background] Nuttall NM, Slade GD, Sanders AE, Steele JG, Allen PF, Lahti S. An empirically derived population-response model of the short form of the Oral Health Impact Profile. Community Dent Oral Epidemiol. 2006 Feb;34(1):18-24. doi: 10.1111/j.1600-0528.2006.00262.x. PMID 16423027
- [Background] Palomares NB, Celeste RK, Oliveira BH, Miguel JA. How does orthodontic treatment affect young adults' oral health-related quality of life? Am J Orthod Dentofacial Orthop. 2012 Jun;141(6):751-8. doi: 10.1016/j.ajodo.2012.01.015. PMID 22640677
- [Background] Ram S, Kumar S, Navazesh M. Management of xerostomia and salivary gland hypofunction. J Calif Dent Assoc. 2011 Sep;39(9):656-9. PMID 22034800
- [Background] Roy EA, Hollins M, Maixner W. Reduction of TMD pain by high-frequency vibration: a spatial and temporal analysis. Pain. 2003 Feb;101(3):267-274. doi: 10.1016/S0304-3959(02)00332-9. PMID 12583869
- [Background] Schulte W, d'Hoedt B, Lukas D, Maunz M, Steppeler M. Periotest for measuring periodontal characteristics--correlation with periodontal bone loss. J Periodontal Res. 1992 May;27(3):184-90. doi: 10.1111/j.1600-0765.1992.tb01667.x. PMID 1608031
- [Background] Schulte W, Lukas D. The Periotest method. Int Dent J. 1992 Dec;42(6):433-40. PMID 1286926
- [Background] Sekhavat AR, Mousavizadeh K, Pakshir HR, Aslani FS. Effect of misoprostol, a prostaglandin E1 analog, on orthodontic tooth movement in rats. Am J Orthod Dentofacial Orthop. 2002 Nov;122(5):542-7. doi: 10.1067/mod.2002.126153. PMID 12439483
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Slade GD. Assessing change in quality of life using the Oral Health Impact Profile. Community Dent Oral Epidemiol. 1998 Feb;26(1):52-61. doi: 10.1111/j.1600-0528.1998.tb02084.x. PMID 9511843
- [Background] Slade GD, Reisine ST. The child oral health impact profile: current status and future directions. Community Dent Oral Epidemiol. 2007 Aug;35 Suppl 1:50-3. doi: 10.1111/j.1600-0528.2007.00405.x. No abstract available. PMID 17615050
- [Background] Sutinen S, Lahti S, Nuttall NM, Sanders AE, Steele JG, Allen PF, Slade GD. Effect of a 1-month vs. a 12-month reference period on responses to the 14-item Oral Health Impact Profile. Eur J Oral Sci. 2007 Jun;115(3):246-9. doi: 10.1111/j.1600-0722.2007.00442.x. PMID 17587301
- [Background] Takahashi I, Nishimura M, Onodera K, Bae JW, Mitani H, Okazaki M, Sasano Y, Mitani H. Expression of MMP-8 and MMP-13 genes in the periodontal ligament during tooth movement in rats. J Dent Res. 2003 Aug;82(8):646-51. doi: 10.1177/154405910308200815. PMID 12885852
- [Background] Tatarakis N, Kinney JS, Inglehart M, Braun TM, Shelburne C, Lang NP, Giannobile WV, Oh TJ. Clinical, microbiological, and salivary biomarker profiles of dental implant patients with type 2 diabetes. Clin Oral Implants Res. 2014 Jul;25(7):803-12. doi: 10.1111/clr.12139. Epub 2013 Feb 27. PMID 23445216
- [Background] Tecco S, D'Attilio M, Tete S, Festa F. Prevalence and type of pain during conventional and self-ligating orthodontic treatment. Eur J Orthod. 2009 Aug;31(4):380-4. doi: 10.1093/ejo/cjp003. Epub 2009 May 22. PMID 19465738
- [Background] Tecco S, Tete S, Perillo L, Chimenti C, Festa F. Maxillary arch width changes during orthodontic treatment with fixed self-ligating and traditional straight-wire appliances. World J Orthod. 2009 Winter;10(4):290-4. PMID 20072744
- [Background] Umesan UK, Chua KL, Krishnan V. Assessing salivary biomarkers for analyzing orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2013 Apr;143(4):446-7. doi: 10.1016/j.ajodo.2013.02.006. No abstract available. PMID 23561400
- [Background] Vs K, K P, Ramesh M, Venkatesan V. The association of serum osteocalcin with the bone mineral density in post menopausal women. J Clin Diagn Res. 2013 May;7(5):814-6. doi: 10.7860/JCDR/2013/5370.2946. Epub 2013 Mar 20. PMID 23814717
- [Background] Yu CC, Chen PH, Liou EJ, Huang CS, Chen YR. A Surgery-first approach in surgical-orthodontic treatment of mandibular prognathism--a case report. Chang Gung Med J. 2010 Nov-Dec;33(6):699-705. PMID 21199616
- [Background] Zhang C, Li J, Zhang L, Zhou Y, Hou W, Quan H, Li X, Chen Y, Yu H. Effects of mechanical vibration on proliferation and osteogenic differentiation of human periodontal ligament stem cells. Arch Oral Biol. 2012 Oct;57(10):1395-407. doi: 10.1016/j.archoralbio.2012.04.010. Epub 2012 May 15. PMID 22595622
- [Background] Zhao L, Wu Z, Zhang Y. Low-magnitude mechanical vibration may be applied clinically to promote dental implant osseointegration. Med Hypotheses. 2009 Apr;72(4):451-2. doi: 10.1016/j.mehy.2008.10.023. Epub 2009 Jan 12. PMID 19138829
- [Derived] Reiss S, Chouinard MC, Frias Landa D, Nanda R, Chandhoke T, Sobue T, Allareddy V, Kuo CL, Mu J, Uribe F. Biomarkers of orthodontic tooth movement with fixed appliances and vibration appliance therapy: a pilot study. Eur J Orthod. 2020 Sep 11;42(4):378-386. doi: 10.1093/ejo/cjaa026. PMID 32572439

RESULTS

PARTICIPANT FLOW:
Groups:
- No Vibration Device+Fixed Appliance Tx: Male and female subjects will randomly assigned to this group to receive fixed appliance orthodontic treatment only. No vibration appliance will be utilized by these patients.
Period: Overall Study
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
Started | 20 | 20
Completed | 20 | 17
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Vibration Device+Fixed Appliance Tx: Subjects will randomly assigned to this group to receive fixed appliance orthodontic treatment in conjunction with vibration therapy (daily use of OrthoAccel Aura device for 20 minutes/day) during the study period.
  Vibration Device: Subjects receiving the OrthoAccel Aura device will be instructed to use the device for 20 minutes/day per the manufacturer's instructions during the study period.
- No Vibration Device+Fixed Appliance Tx+Female: Subjects will randomly assigned to this group to receive fixed appliance orthodontic treatment only and no vibration treatment.
- Total: Total of all reporting groups
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx+Female | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (5.8) | 19.7 (5.5) | 20.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Expression of Salivary Biomarkers of Bone Remodeling
Description: Saliva will be collected as T0 (Baseline), T1 (5-6 weeks), T2 (10-12 weeks), T3 (15-17 weeks). Saliva will be analysed for a variety of biomarkers with protein quantified by ELISA assay at each time point for each subject.
Time Frame: Up to Week 17 of alignment (From T0 to T3)
Population: Vibration and Control subjects-- all subjects in the study averaged across all time points per group.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- No Vibration Device+Fixed Appliance Tx: Male and female subjects will randomly assigned to this group to receive fixed appliance orthodontic treatment in conjunction with vibration therapy (daily use of OrthoAccel Aura device for 20 minutes/day) during the study period.
  Vibration Device: Subjects receiving the OrthoAccel Aura device will be instructed to use the device for 20 minutes/day per the manufacturer's instructions during the study period.
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
Number analyzed (Participants) | 20 | 20
pg/mL
  TNFa | -1.62 (8.73) | 0.5 (13.72)
  IL-6 | -1.95 (8.03) | 0.47 (11.09)
  MMP-9 | -17957.59 (71966.29) | 6783.71 (18101.55)
  IL-3 | -0.52 (48.39) | -1.6 (22.85)
  IL-8 | -35.53 (175.65) | -78.66 (347.4)
  DKK-1 | -7.39 (115.65) | -14.7 (62.17)
  MMP-13 | -20.27 (94.22) | -2.27 (39.37)
  SOST | -1.71 (8.25) | 1.53 (4.82)
  RANKL | 9.28 (49.59) | 2.59 (33.46)
  OPN | -371.93 (1991.37) | 134.44 (2973.88)
  IL-11 | -90.87 (423.73) | 46.15 (485.07)
  IL-18 | -3.46 (15.79) | -0.35 (4.81)
  OPG | -2.69 (62.90) | 21.05 (103.62)
  TGF-B1 | 0.68 (3.46) | -9.49 (36.82)

2. Primary Outcome: Alignment of Mandibular Anterior Teeth
Description: At each study visit, alginate impressions will be taken on each subject. These models will be analyzed by 2 examiners to calculate the alignment based on Little's Irregularity Index. Measure Description: Little's Irregularity index measures the interproximal contact displacement in mm between the anterior teeth segment from the mesial of the canine on one side to the mesial aspect of the contralateral canine.
Time Frame: Up to Week 17
Population: All subjects (40 total)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
Number analyzed (Participants) | 20 | 20
mm | 6.49 (3.43) | 7.47 (3.62)

3. Secondary Outcome: Tooth Mobility
Description: The degree of tooth mobility will be used using a Periotest device (Siemens, Bensheim, Germany) on the central incisors, canines and 2nd premolars in both mandibular quadrants as previously described by Liou et al. The archwire will be removed and the Periotest measurements will be taken in triplicate, with means recorded. The Periotest's scale ranges from -8 to +50. The lower the Periotest value, the higher is the stability / damping effect of the test object (tooth or implant). -8 to 0 indicates high stability with minimal movement, +1-+9 indicates some degree of mobility (moderate) and +10 to +50 indicates severe mobility.
Time Frame: Up to Week 17
Population: All subjects (40 total).
Measure: Mean (Standard Deviation); unit: PTV
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
Number analyzed (Participants) | 20 | 20
PTV | 2.34 (1.10) | 2.42 (0.69)

4. Secondary Outcome: Orthodontic Pain Assessment
Description: Subjects will be given a pain diary on the baseline (T0), visits T1 & T2 to record the level of orthodontic pain each evening for the first 7 days after each study visit. The degree of pain was assessed using a metric Visual Analog Scale. The patient was given a scale that was a 100 mm in length. At 0 mm on the scale line, the pain level would be "0" indicating no pain. At the higher end of the line scale (the 100 mm mark), the pain level was considered the most severe. Data presented here indicates the mean VAS scores in mm for the 1st week following each study visit. The average values indicate the measure along the scale.
Time Frame: Up to Week 17
Population: All subjects (40 total).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
Number analyzed (Participants) | 20 | 20
mm
  T0 | 33.11 (25.19) | 35.25 (22.46)
  T1 | 13.92 (18.17) | 14.4 (16.42)
  T2 | 24.12 (23.3) | 27.66 (24.09)

5. Secondary Outcome: Oral Health Quality of Life
Description: To assess the impact of the vibration appliance on the overall oral health quality of life of the subject, subjects will be given an Oral Health Impact Profile (OHIP-14) questionnaire. The OHIP-14 consists of 14 question areas divided into specific dimensions including functional limitation, physical pain, psychological discomfort, physical disability, psychological and social disability and overall life handicap from orthodontic treatment with or without the vibration appliance. For the OHIP questionnaire, responses are coded 0 (never or not applicable), 1 (hardly ever), 2 (occasionally), 3 (fairly often) or 4 (very often). As a general rule, the greater the OHIP score, the more of an impact a particular intervention had on the patient's overall quality of life. The scores for the overall OHIP-14 range from 0-56, with values closer to 0 indicating minimal impact on quality of life and values closer to 56 indicating great impact on quality of life.
Time Frame: Up to Week 17
Population: All subjects (40 total).
Measure: Mean (Standard Deviation); unit: Units on OHIP-14 Scale
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
Number analyzed (Participants) | 20 | 20
Units on OHIP-14 Scale
  T0 | 4.5 (3.71) | 5.94 (3.74)
  T1 | 5.56 (3.73) | 6.12 (3.36)
  T2 | 4.4 (3.96) | 4.91 (3.54)
  T3 | 3.27 (2.8) | 3.9 (2.79)

ADVERSE EVENTS:
Time Frame: For each subject up to 17 weeks of their participation in the study.
Description: Adverse Event Reporting was conducting in accordance with the Institutional Review Board (IRB) protocol at the University of Connecticut Health Center (14-117-2). Adverse event data collected systematically per set times in subject recruitment. During the study, there were a total of 6 meetings.
Arm/Group | Vibration Device+Fixed Appliance Tx | No Vibration Device+Fixed Appliance Tx
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT02119455/Prot_SAP_000.pdf